CLINICAL TRIAL: NCT07363239
Title: A New Concept of Safety Distance to Place Implants in the Area of the Inferior Alveolar Canal to Avoid Neurosensory Disturbance: A Retrospective CBCT Study
Brief Title: CBCT-Based Safety Distance for Implant Placement Near the Inferior Alveolar Canal
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ghada Adayil, Lecturer, Faculty of Dentistry, Cairo University, Cairo University
Other Study IDs: 12/25
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Inferior Alveolar Approximation; Implants
Keywords: inferior alveolar nerve; implants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- implants placed more than 2mm from the inferior alveolar canal
  Interventions: Other: nerve approximation group
- Implant proximity < 2 mm

INTERVENTIONS:
Other: nerve approximation group — implants placed with distance more than 2 mm from the inferior alveolar canal
  Groups: implants placed more than 2mm from the inferior alveolar canal

SUMMARY:
o evaluate the radiologic proximity of mandibular dental implants placed less than 2 mm from the inferior alveolar canal using cone-beam computed tomography (CBCT), and to determine the relationship between implant-canal distance and the occurrence of postoperative neurosensory disturbances.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 21 years.
2. Implants placed in mandibular first/second premolar or molar positions (Froum et al., 2021).
3. Patients without neurosensory changes following implant placement and healing (Froum et al., 2021).
4. Patients with neurosensory changes after implant placement, including paresthesia, anesthesia, dysesthesia (and neuralgia where applicable) (Froum et al., 2021).

Exclusion Criteria:

1. Incomplete records preventing outcome ascertainment (Froum et al., 2021).
2. Refusal/unavailability of postoperative CBCT when clinically required for evaluation (Froum et al., 2021).
3. Poor-quality CBCT scans or scatter artifacts interfering with evaluation (Froum et al., 2021).
4. Contraindications for radiographs (e.g., pregnancy/breastfeeding) in cases where additional imaging would otherwise be clinically required (Froum et al., 2021).
5. Implants placed after mental foramen

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consisted of adult patients with available CBCT scans, retrospectively evaluated for implant-related anatomical assessment in the region of the inferior alveolar canal.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-01-25 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Neurosensory outcome | 6 months
  presence/absence of neurosensory changes after implant placement, classified as reported in records (none, paresthesia, anesthesia, dysesthesia, neuralgia)